CLINICAL TRIAL: NCT04040166
Title: PET/MR of the Carotid Arteries With 68Ga DOTATATE in Patients Following Head and Neck Radiation Therapy and at Risk of Cerebrovascular Events
Brief Title: Carotid PET/MRI With DOTATATE in Patients Post Head and Neck Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-6313
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Head & Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Carotid PET/MRI With DOTATATE in patients post head and neck radiation therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MRI scan with 68Ga DOTATATE (Other): PET/MRI scan with 68Ga DOTATATE of carotid arteries in in patients following head and neck radiation therapy
  Interventions: Diagnostic Test: PET/MRI of carotid arteries with 68Ga DOTATATE

INTERVENTIONS:
Diagnostic Test: PET/MRI of carotid arteries with 68Ga DOTATATE — PET/MRI of carotid arteries with 68Ga DOTATATE in patients post head and neck radiation therapy

SUMMARY:
The improvement of comprehensive multi-modality treatment and radiotherapy (RT) technology has resulted in an improved survival rate of head and neck malignancies within recent decades. As survival increases, late toxicity from cancer therapy becomes a larger burden. Radiation induced vascular injury following RT is a recognized complication of radiotherapy. Diagnosis of vascular changes predominately relies on non-invasive imaging techniques. Doppler ultrasound assessment has been proven as a good indicator of diffuse atherosclerotic disease and a significant predictor of future vascular events. New opportunities are provided by the recent introduction of the hybrid PET/MRI scanners for investigating the synergistic effect of these two modalities without the challenge of image co-registration. It has been shown that the PET system integrated with the MRI scanner performs the same as the PET portion of a PET/CT for various cancers and cardiovascular indications. MRI allows better delineation of the carotid artery and atherosclerotic plaque when compared with CT due to the superior soft tissue contrast. The PET/MRI system acquires the PET and MRI simultaneously allowing for perfect alignment between the 2 sets of images, when compared with the sequential acquisition in PET/CT where minor head movements can cause misalignment. There is evidence in the literature that 68-Ga DOTA-TATE PET-imaging can serve as a surrogate marker for evidence of invasion into the vessel wall and thereby possibly detects early, developing atherosclerotic plaque. Thus, combined PET and MR with 68-Ga DOTA-TATE should be a promising imaging tool to screen and characterize patients at risk for radiation induced carotid injury.

In this study, DOTATATE-PET/MR will be performed in up to 60 patients with a history of radiation therapy for head and neck squamous cell carcinoma over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* previously treated with radiation for head and neck malignancy;
* Age Group: ≥30 years;
* Patients who have no contraindications to PET/MRI;
* No allergy to contrast agents.

Exclusion Criteria:

* Pregnant females;
* Age group: < 30 years;
* Allergy to MR contrast agents;
* Pacemakers/ICD/Claustrophobic patients.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Validity of PET/MRI with 68Ga DOTATATE of carotid arteries | complete of enrollment, an average of two years
  Macrophage activity detected by 68Ga DOTATATE PET/MRI of carotid arteries in patients at risk for vascular events post radiation of head and neck squamous cell carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada